CLINICAL TRIAL: NCT01491009
Title: Comparison of Remifentanil With Dexmedetomidine or Midazolam in Regards of Sedation Effectivity and Postoperative Cognitive Functions in Cystoscopies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayşe Hande Arpacı, Dr. at Department of Anaesthesiology and Reanimation, Gazi University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-154
Record Dates: First submitted 2011-12-06; First posted 2011-12-13 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Postoperative Cognitive Functions
Keywords: Dexmedetomidine; midazolam; remifentanil; mini-mental state examination; monitored anaesthesia care; cystoscopy; sedation
MeSH Terms: interventions — Remifentanil; Midazolam

INTERVENTIONS:
Drug: Remifentanil — IV infusion
Drug: Midazolam — IV infusion

SUMMARY:
The aim of the study was to compare the effects of remifentanil-dexmedetomidine and remifentanil-midazolam with mini-mental state examination (MMSE) in monitored anesthesia care (MAC) patients undergoing cystoscopy.

DETAILED DESCRIPTION:
Forty patients undergoing cystoscopy receiving remifentanil infusion of 0.05 microgram per kg-1 min-1 were randomized into two groups: Either dexmedetomidine 1 microgram per kg -1 (GroupD) or midazolam 0.2 mg kg-1h-1 (GroupM) were administered intravenously for the first 10 minutes. Subsequently anesthesia was maintained by using the bispectral index(BIS) as a continuous infusion of dexmedetomidine 0.2-0.7 microgram per kg-1h-1 or midazolam 0.05-0.15 mgkg-1h-1. Heart rate, mean arterial pressure, MMSE, sedation and the patient's and surgeon's satisfaction were determined.

ELIGIBILITY:
Inclusion Criteria:

* patients with indication of cystoscopy must be able to have sedation

Exclusion Criteria:

* hypersensitivity to drugs used
* morbid obesity
* coronary disease
* diabetes mellitus and other endocrinologic diseases
* pregnancy
* psychomotor diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2007-02 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Degree of sedative efficiency | During cystoscopy procedure
  Bispectral Index (BIS) was used.
Degree of cognitive functions | Postoperative 60 minutes
  mini-mental state examination(MMSE) test was used.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Arpacı, M.D., Principal Investigator — Gazi University; Füsun Bozkırlı, M.D., Study Director — Gazi University
Locations (1):
- Gazi University Faculty of Medicine Hospital, Ankara, Turkey (Türkiye)